CLINICAL TRIAL: NCT05344196
Title: Examining the Effect of a Novel Stress Reduction Intervention no the Control of Prediabetes: A Feasibility Study
Brief Title: Emotional Awareness and Expression Therapy for Prediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Mark A. Lumley, Professor, Wayne State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-19-09-1275
Record Dates: First submitted 2022-04-07; First posted 2022-04-25 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: PreDiabetes
Keywords: Stress reduction; Emotional Awareness and Expression Therapy
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Intervention Model Description: Several cohorts of people with prediabetes will be given the treatment and tracked with respect to outcomes from before to after treatment and follow-up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified EAET for Prediabetes (Experimental): Small groups of people with prediabetes will meet for 4, weekly, 2-hour sessions by telehealth, and will engage in modified EAET for prediabetes
  Interventions: Behavioral: Modified EAET for prediabetes

INTERVENTIONS:
Behavioral: Modified EAET for prediabetes — Attempts to reduce stress and improve health behavior by engaging in emotional awareness and expression leading to changes in interpersonal relationships and health behavior

SUMMARY:
This feasibility study seeks to develop and pilot test Emotional Awareness and Expression Therapy as a possible treatment for people with prediabetes.

DETAILED DESCRIPTION:
Prediabetes is a clinical condition in which hemoglobin A1C is between 5.6 and 6.4, and is usually associated with being overweight, poor diet, limited exercise, and psychological stress. This condition develops in to Type II diabetes in many people, and interventions to prevent such progression are needed. Because stress can directly negative impact blood glucose metabolism and can indirectly affect it through unhealthy behaviors (e.g., diet, exercise), it may be possible to reduce stress and improve clinical outcomes. Although most stress management approaches help people to calm their physiology and reduce their negative emotions, another approach to stress treatment is to help people disclose emotionally difficult experiences, become aware of and express their emotions, and change interpersonal relationships by becoming more assertive as well as more open/connected.

Emotional Awareness and Expression Therapy (EAET) is an approach to stress reduction that uses these principles and it has been shown to be effective for somatic symptom disorders like chronic pain. In this study, we will adapt EAET to the prediabetes context and test its feasibility, acceptability and initial efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated with Wayne State University (faculty, staff, student, or family member/friend thereof)
* HbA1C value of 5.7% to 6.4%
* overweight or obese (≥25 kg/m2) Also, if over ≥ 18 and < 45 years of age must have at least one of the following: a) physical inactivity, b) close family history of diabetes, c) history of hyperlipidemia, d) history of hypertension, e) history of gestational diabetes, and/or f) from high risk race groups (e.g., African American, Latino, Native American, and pacific Islander).

Exclusion Criteria:

* Confirmed history of Type 2 Diabetes
* have prediabetes being treated pharmacologically
* pregnant
* taking medications that affect blood glucose (e.g., corticosteroids)
* chronic depression or major psychotic disorder
* any comorbidities that limit survival or ability to tolerate the intervention (Cushing's, cancer treatment, asthma with inhaled corticosteroids, unstable CAD or MI in last 6 months, CHF, COPD requiring oxygen, chronic kidney disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
HbA1c | Change from baseline to 3-month follow-up and 6-month follow-up
  Hemoglobin A1c from venous blood
C-peptide | Change from baseline to 3-month follow-up and 6-month follow-up
  venous blood surrogate marker of insulin levels

SECONDARY OUTCOMES:
Perceived Stress Scale | Change from baseline to 3-month follow-up and 6-month follow-up
  Psychological stress (scores from 0 to 40; higher scores indicate more perceived stress)
Body mass index | Change from baseline to 3-month follow-up and 6-month follow-up
  Measure of overweight / obesity
Health behavior | Change from baseline to 3-month follow-up and 6-month follow-up
  Self-reported exercise and diet over the past week

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No